CLINICAL TRIAL: NCT02875496
Title: Reference Database & Longitudinal Registry of the Normal and Pathological Aging Brain: Brain Network Activation Analysis (BNA™) for the Adult and Elderly Population Using Evoked Response Potentials
Brief Title: Reference Database & Longitudinal Registry of the Normal and Pathological Aging Brain
Acronym: (BNA™)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-26
Record Dates: First submitted 2016-08-04; First posted 2016-08-23 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Early Onset Alzheimer Disease; Mild Cognitive Impairment; Depression; Aging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy aging: Subjects meeting criteria for healthy aging No intervention administered
- Early Alzheimer Disease: Subjects meeting criteria for Early Alzheimer Disease No intervention administered
- Depression: Subjects meeting criteria for Depression No intervention administered
- MCI-Mild Cognitive Impairment: Subjects meeting criteria for MCI-Mild Cognitive Impairment No intervention administered
- General Arm: Subjects not meeting criteria for any of the other arms (Healthy, Early Alzheimer's, Depression, or MCI)

SUMMARY:
Establishment of a BNA reference database for the Adult and Elderly Population. Hypothesis-generating study designed to collect data that will aid in future scientific and engineering exploration of correlations between clinical assessments and BNA scores. The results are primarily intended for scientific inquiry and engineering development purposes, and may be used in future regulatory submissions.

DETAILED DESCRIPTION:
Currently, there is no reliable, bedside, and non-invasive method for assessing connectivity changes in electrophysiological activity of the brain associated with brain-related pathologies, e.g., concussion, ADHD, autistic spectrum disorders (ASD), etc. Event Related Potentials (ERPs), which are temporal reflections of the neural mass electrical activity of cells in specific regions of the brain that occur in response to stimuli, may offer such a method, as they provide both a non-invasive and portable measure of brain function. The ERPs provide excellent temporal information, but spatial resolution for ERPs has traditionally been limited. However, by using high-density electroencephalograph (EEG) recording, spatial resolution for ERPs is improved significantly. The paradigm for the current study will combine neurophysiological knowledge with mathematical signal processing and pattern recognition methods (BNA) to temporally and spatially map brain function, connectivity and synchronization.

The need of objective measures that will help the clinician in its decision-making in brain-related pathologies is recognized. BNA is a new imaging modality that has been developed to fill this gap.

ELIGIBILITY:
For ALL arms:

Inclusion Criteria:

* Currently resides in The Villages community
* Age 50-years and above.
* Able to speak, read and understand English
* Willingness to participate and able to give informed consent.
* If corrected vision: only Glasses should be used during the study testing

Exclusion Criteria:

* Currently with lice or open wounds on scalp.
* Any CNS neurologic disorder
* Significant sensory deficits.
* Use of a hearing aid that occupies the ear canal
* Any neuropsychological disorders
* History of special education
* Substance abuse in the last 3 months
* History of any clinically significant brain trauma as determined by the investigator.
* Clinically diagnosed with a concussion in the past year.

For Arm 1 Healthy

Inclusion Criteria:

* BDI score <14
* Subjects Not meeting diagnostic criteria for MDD per the DSM IV-TR,
* MMSE score ≥25

Exclusion Criteria:

* Any chronic disease or condition which affects the nervous system as determined by clinical neurological evaluation, medical history or PI discretion.
* Any psychiatric disorder,
* History of any medication affecting CNS within the last 3 months

For Arm 2 Early Alzheimer's Disease

Inclusion Criteria:

* BDI score <14
* Subjects Not meeting diagnostic criteria for MDD per the DSM IV-TR, as determined by clinical evaluation by a research clinician and the Mini International Neuropsychiatric Interview (MINI).
* MMSE score <24
* MoCA<20
* Presence of an early and significant episodic memory impairment

Exclusion Criteria:

* Any chronic disease or condition other than current pathology
* Any other psychiatric disorder
* CNS medications within the short period of time prior to the EEG testing which are not in a medically stable treatment phase.

For Arm 3 Depression

Inclusion Criteria:

* BDI score >14
* Subjects meeting full diagnostic criteria for MDD without psychotic features per the DSM IV-TR
* HAM-D 17-item: Total score of 16 or higher at visit 1.

Exclusion Criteria:

* Any chronic disease or condition other than current pathology
* Any psychiatric disorder other than Depression
* CNS medications within the short period of time prior to the EEG testing which are not in a medically stable treatment phase.

For Arm 4 Mild Cognitive Impairment

Inclusion Criteria:

* BDI score <14
* Subjects Not meeting diagnostic criteria for MDD per the DSM IV-TR
* MMSE scores according to Number of years of Education:

MMSE score Years of Education 17-18 ≤6 20-21 7-8 23-24 ≥10

-20<MoCA score >26

Exclusion Criteria:

* Any chronic disease or condition other than current pathology
* Any other psychiatric disorder
* CNS medications within the short period of time prior to the EEG testing which are not in a medically stable treatment phase.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 2000 subjects, from both genders, aged 50- years and above will be recruited and stratified to age groups. Once enrollment reaches the below numbers for each age group, subjects will be statistically stratified and analyzed in 4 different Arms, one Normative and three Pathologies, according to a prospective statistical plan and based on the prevalence of common pathological conditions in each age group; this will be determined by analysis of the literature, analysis of study demographics and concomitant diseases, and on the PI and/or sponsor's discretion. Suggested enrollment numbers for the different age groups and different Arms are:
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-08; Primary Completion 2022-08 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Developing a BNA database for healthy aging population. | 2 years
  Functional networks of brain activity in healthy aging individuals measured using analysis of EEG Event Related Potential (ERP) data Clinical assessments battery will be utilized in order to establish different sets of BNA database for age related pathology and healthy aging.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lowenkron, MD, Principal Investigator — Chief Medical Officer, The Villages Health; Carla VandeWeerd, PhD, Principal Investigator — Director of Research, The Villages Health
Locations (1):
- The Villages Health, The Villages, Florida, United States

IPD SHARING:
Plan to Share IPD: No